CLINICAL TRIAL: NCT03766360
Title: A Social Functioning Intervention to Target Depression Post Bariatric Surgery
Brief Title: Bariatric Surgery Study
Acronym: SIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jonathan Kanter, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005196
Record Dates: First submitted 2018-11-27; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Depression; Quality of Life; Interpersonal Relations
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAP Intervention Group (Experimental): All of the clients in the FAP intervention group will begin treatment at the same time and complete 3 assessments.
  Interventions: Behavioral: Functional Analytical Psychotherapy (FAP)
- Control Group (No Intervention): The clients in the control group will take their assessments at the same time as those in the FAP intervention group.

INTERVENTIONS:
Behavioral: Functional Analytical Psychotherapy (FAP) — The intervention itself is based on the procedures of Functional Analytic Psychotherapy, a behavioral intervention focusing on improving social functioning.
  Arms: FAP Intervention Group

SUMMARY:
The current study proposes an open clinical trial to investigate the effectiveness of a social functioning intervention on bariatric surgery outcomes and depression. The treatment will be administered in a group format over 10 weekly/biweekly sessions and will take place at the University of Washington Weight Loss Management Clinic (WLMC) at the Roosevelt Clinic location. Effects of the intervention will be measured with self-report questionnaires and by self-report of behaviors outside of assessment sessions (via questionnaires and self-report of adherence to treatment). Data collection will occur at specific time points including before treatment, after treatment, and two months after treatment.

DETAILED DESCRIPTION:
As of 2009, 344,000 bariatric procedures were performed annually . Although some studies report depressive symptoms decrease in the 6 months after bariatric surgery, there is growing body of literature suggesting there exists a subgroup of patients whose depressive symptoms worsen after surgery and the likelihood of developing depressive symptoms increases longitudinally. Depression can be an indicator of an increased risk of self-harm and additional studies have found that the risk of suicide may increase post bariatric surgery compared to obese individuals who have not undergone surgery.

Research supports that psychosocial factors contribute to successful postoperative outcomes. Functional Analytic Psychotherapy shows potential to impact social variables that may be relevant to bariatric surgery outcomes including depression. In this context, FAP aims to improve interpersonal relationships through experientially teaching skills intended to increase social connection. FAP also seeks to increase awareness, which includes the ability to view interpersonal interactions from multiple perspectives, allowing new interpersonal skills to emerge.

The present study seeks to evaluate the use of a FAP group to enhance interpersonal relating with a sample of post-bariatric surgery patients. Measures will be collected on quality of life and variables involved in interpersonal connectedness.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Speak English as a primary language
* Had Bariatric Surgery in the past 6-24 months (bypasses (Roux-en-Y) or sleeves)
* Yes to one or both of the first two PHQ-9 Questions
* Not pregnant
* Not traveling anywhere in the next 6 months
* No surgeries scheduled in the next 12 months

Exclusion Criteria:

• No exclusion criteria are utilized in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  based directly on the nine diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Diploma in Social Medicine-IV
Patient Health Questionnaire-9 (PHQ-9) | Post Intervention (Approximately 12 Weeks from Baseline)
  based directly on the nine diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Diploma in Social Medicine-IV
Patient Health Questionnaire-9 (PHQ-9) | Follow Up (3 Months after Intervention)
  based directly on the nine diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Diploma in Social Medicine-IV

SECONDARY OUTCOMES:
World Health Organization Quality of Life | Baseline
  a measure of an individual's physical health, psychological state, personal beliefs, social relationships and their relationship to salient features of their environment.
World Health Organization Quality of Life | Post Intervention (Approximately 12 Weeks from Baseline)
  a measure of an individual's physical health, psychological state, personal beliefs, social relationships and their relationship to salient features of their environment.
World Health Organization Quality of Life | Follow Up (3 Months after Intervention)
  a measure of an individual's physical health, psychological state, personal beliefs, social relationships and their relationship to salient features of their environment.
Drug Abuse Screening Test | Baseline
  a sensitive screening instrument for the abuse of drugs other than alcohol
Drug Abuse Screening Test | Post Intervention (Approximately 12 Weeks from Baseline)
  a sensitive screening instrument for the abuse of drugs other than alcohol
Drug Abuse Screening Test | Follow Up (3 Months after Intervention)
  a sensitive screening instrument for the abuse of drugs other than alcohol
Paffenbarger Physical Activity Questionnaire | Baseline
  asks participants about their current and previous exercise habits
Paffenbarger Physical Activity Questionnaire | Post Intervention (Approximately 12 Weeks from Baseline)
  asks participants about their current and previous exercise habits
Paffenbarger Physical Activity Questionnaire | Follow Up (3 Months after Intervention)
  asks participants about their current and previous exercise habits
Proximal Change Variables | Baseline
  assesses participant's eating habits as well as tobacco and alcohol use
Proximal Change Variables | Post Intervention (Approximately 12 Weeks from Baseline)
  assesses participant's eating habits as well as tobacco and alcohol use
Proximal Change Variables | Follow Up (3 Months after Intervention)
  assesses participant's eating habits as well as tobacco and alcohol use
Weight Control Questionnaire | Baseline
  asks participants to report if they have ever used any weight control practices
Weight Control Questionnaire | Post Intervention (Approximately 12 Weeks from Baseline)
  asks participants to report if they have ever used any weight control practices
Weight Control Questionnaire | Follow Up (3 Months after Intervention)
  asks participants to report if they have ever used any weight control practices
Fear of Intimacy Scale (FIS) | Baseline
  The FIS is a 35 item measure of self-disclosure, social intimacy, and social desirability. All items are scored on a 5-point Likert scale
Fear of Intimacy Scale (FIS) | Post Intervention (Approximately 12 Weeks from Baseline)
  The FIS is a 35 item measure of self-disclosure, social intimacy, and social desirability. All items are scored on a 5-point Likert scale
Fear of Intimacy Scale (FIS) | Follow Up (3 Months after Intervention)
  The FIS is a 35 item measure of self-disclosure, social intimacy, and social desirability. All items are scored on a 5-point Likert scale
Social Support Survey | Baseline
  provides an assessment of several domains of social support including tangible support, emotional support, affective support, and positive support
Social Support Survey | Post Intervention (Approximately 12 Weeks from Baseline)
  provides an assessment of several domains of social support including tangible support, emotional support, affective support, and positive support
Social Support Survey | Follow Up (3 Months after Intervention)
  provides an assessment of several domains of social support including tangible support, emotional support, affective support, and positive support
University of California, Los Angeles Loneliness Scale | Baseline
  designed to measure one's subjective feelings of loneliness as well as feelings of social isolation
University of California, Los Angeles Loneliness Scale | Post Intervention (Approximately 12 Weeks from Baseline)
  designed to measure one's subjective feelings of loneliness as well as feelings of social isolation
University of California, Los Angeles Loneliness Scale | Follow Up (3 Months after Intervention)
  designed to measure one's subjective feelings of loneliness as well as feelings of social isolation

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Loss Management Center at UWMC-Roosevelt, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Switzer, N.J., Debru, E., Church, N. et al. Curr Cardiovasc Risk Rep (2016) 10: 12. https://doi.org/10.1007/s12170-016-0492-7
- [Background] Mitchell JE, Crosby R, de Zwaan M, Engel S, Roerig J, Steffen K, Gordon KH, Karr T, Lavender J, Wonderlich S. Possible risk factors for increased suicide following bariatric surgery. Obesity (Silver Spring). 2013 Apr;21(4):665-72. doi: 10.1002/oby.20066. PMID 23404774
- [Background] Sarwer DB, Moore RH, Spitzer JC, Wadden TA, Raper SE, Williams NN. A pilot study investigating the efficacy of postoperative dietary counseling to improve outcomes after bariatric surgery. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):561-8. doi: 10.1016/j.soard.2012.02.010. Epub 2012 Mar 21. PMID 22551576
- [Background] Kohlenberg, R. J., & Tsai, M. (1991). Functional analytic psychotherapy: Creating intense and curative therapeutic relationships. New York, NY, US: Plenum Press. http://dx.doi.org/10.1007/978-0-387-70855-3